CLINICAL TRIAL: NCT05226442
Title: A Prospective Randomized Pilot Trial on Safety and Feasibility of Argatroban As Anticoagulant in Patients with Extracorporeal Membrane Oxygenation (ECMO)
Brief Title: Safety and Feasibility of Argatroban As Anticoagulant in Adults with ECMO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Thomas Staudinger, Prof., MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Argatroban_ECMO
Record Dates: First submitted 2021-12-04; First posted 2022-02-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Extracorporeal Membrane Oxygenation Complication; Anticoagulants and Bleeding Disorders
MeSH Terms: conditions — Hemostatic Disorders | interventions — argatroban; Heparin

STUDY DESIGN:
Intervention Model Description: Randomization ratio of 1:1 for anticoagulation with Argatroban or Unfractionated Heparin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Argatroban (Experimental): Continuous infusion of 0,3μg/kg/min to target an aPTT of 50-70sec and/or Hemoclot of 0,60 - 0,80 µg/mL
  Interventions: Drug: Argatroban
- Unfractionated Heparin (Active Comparator): Continuous infusion of Unfractionated Heparin to target an aPTT of 50-60 seconds and/or Anti-Xa level between 0.20 and 0.30 IU/ml and/or thrombin time >20sec.
  Interventions: Drug: Unfractionated heparin

INTERVENTIONS:
Drug: Argatroban — Argatroban is a synthetic, univalent DTI, that directly binds to the catalytic thrombin binding site exerting its effects
  Arms: Argatroban
Drug: Unfractionated heparin — Unfractionated heparin produces its major anticoagulant effect by inactivating thrombin and activated factor X (factor Xa) through an antithrombin (AT)-dependent mechanism.
  Arms: Unfractionated Heparin

SUMMARY:
This prospective, randomized, controlled pilot trial aims to assess the safety and feasibility of Argatroban as an alternative anticoagulant to unfractionated heparin in patients receiving extracorporeal membrane oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Minimum Age 18 years
* VV- or VA-ECMO therapy
* Minimum of 24h planned ECMO-therapy

Exclusion Criteria:

* History of Heparin-induced thrombocytopenia (HIT)
* High risk of bleeding, contraindication for anticoagulation (eg. active GI-bleeding, Intracerebral bleeding; Platelet count <50G/l, congenital bleeding disorder)
* Pregnancy
* Severe Liver disease (SOFA score liver domain 4 points = Bilirubin >12mg/dl)
* Postoperative admission
* Strong lupus anticoagulant or acquired intrinsic clotting factor deficiency at admission (APTT >50 sec without anticoagulation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-07-07 (Actual)

PRIMARY OUTCOMES:
Bleeding and thrombosis with Argatroban compared to unfractionated Heparin (UFH) | From date of randomization until the date of ECMO discontinuation, or death, whichever came first, assessed up to 120 days
  Bleeding will be assessed continuously by the investigators according to the BARC bleeding classification, where bleeding type 2 or higher will be considered as clinically significant bleeding; outcome measures will be the incidence of clinically significant bleeding per ECMO day and time to first bleeding; thrombosis is defined as any occurence of thromboembolism including membrane lung exchange due to suspected thrombosis, pulmonary embolism or deep vein thrombosis; outcome measures will be the incidence of thromboembolism per ECMO day and the time to first thromboembolism

SECONDARY OUTCOMES:
study enrollment, study completion and ability to achieve target values of Argatroban as anticoagulant in ECMO | From date of randomization until the date of ECMO discontinuation, or death, whichever came first, assessed up to 120 days
  ratio of screened to included patients, proportion of patients who completed the study according to the protocol, proportion of coagulation tests within range and total number of dose adjustments

OTHER OUTCOMES:
Transfusion rate of packed red blood cells assessed as total units/ECMO day | From date of randomization until the date of ECMO discontinuation, or death, whichever came first, assessed up to 120 days
  Assessment of the total amount of units (250-300ml each) packed red blood cells transfused per ECMO day following a transfusion threshold of Hb<8g/dl
Grading of bleeding | From date of randomization until the date of ECMO discontinuation, or death, whichever came first, assessed up to 120 days
  According to the Bleeding Academic Research Consortium type 1 - 5 (Type 1: Bleeding that is not actionable; Type 2: Any clinically overt sign of hemorrhage that "is actionable" and requires diagnostic studies, hospitalization, or treatment by a health care professional; Type 3a. Overt bleeding plus hemoglobin drop of 3 to < 5 g/dL (provided hemoglobin drop is related to bleed); transfusion with overt bleeding; Type 3b. Overt bleeding plus hemoglobin drop < 5 g/dL (provided hemoglobin drop is related to bleed); cardiac tamponade; bleeding requiring surgical intervention for control; bleeding requiring IV vasoactive agents; type 3c. Intracranial hemorrhage confirmed by autopsy, imaging, or lumbar puncture; intraocular bleed compromising vision; Type 4: CABG-related bleeding within 48 hours; Type 5a. Probable fatal bleeding; Type 5b. Definite fatal bleeding (overt or autopsy or imaging confirmation)
Mortality rate at day 28/90 | Until 90 days after start of study drug administration
  assessed by chart review or telephone call

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Staudinger, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
upon reasonable request